CLINICAL TRIAL: NCT06577168
Title: The Prevalence and Predictors of Menstrual Pattern Within Six Months of Levonogestrel IUS Insertion.
Brief Title: Menstrual Pattern Within Six Months of Levonogestrel IUS Insertion
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mariam Samy Lotfy, Resident doctor, Assiut University
Other Study IDs: Contraception
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Contraception

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Other: Levonogestrel Intrauterine system (LNG-IUS) — Contraception method

SUMMARY:
The purpose of this study is to systematically calculate the mean number of bleeding-only, spotting-only, and bleeding and/or spotting days experienced by a population of reproductive aged,52 mg levonogestrel Intrauterine System(LNG-IUS) users.

DETAILED DESCRIPTION:
The levonogestrel Intrauterine system (LNG-IUS)(52 mg per 20mg per day release) is associated with medically benign changes to the menstrual pattern. Amenorrhea, the complete cessation of vaginal bleeding for at least 90 consecutive days, is perhaps the most extreme bleeding pattern experienced by some users during the first year. Amenorrhea prevalence is positively associated with duration of use, with approximately 8% of users.

ELIGIBILITY:
Inclusion Criteria:

* Included participants with normal regular menses prior to LNG-IUS

insertion

* Included participants of any age, race, ethnicity, or parity
* Contained bleeding and/or spotting data on the 52 mg (20 mg/d) LNG-IUS
* Collected daily menstrual bleeding data from written diaries for at least 90 consecutive days

Exclusion Criteria:

* Heavy or prolonged menstrual bleeding (menorrhagia)
* Actively breastfeeding
* Hormonal long-acting reversible contraceptive method (LNG-IUS, implant) within 3 months of enrollment
* Hormonal injectable contraceptive use within 6 months of enrollment
* First 3 months (90 days) of data from women with postpartum or postabortion LNG-IUS insertions
* Any anatomical or pathological condition (ie, uterine fibroids) that may have an impact on baseline menstrual bleeding pattern

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Females in reproductive age
Study Population: Females at reproductive age (18-45)
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Mean number of days with menstrual bleeding changes | Six months after insertion of levonogestrel Intrauterine system
  This include calculating the average number of days per month with bleeding-only, spotting-only,and bleeding and/or spotting in reproductive aged women using a 52 mg levonogestrel Intrauterine system (LNG-IUS) within the first six months ofuse, according to World Health Organization standards.

CONTACTS AND LOCATIONS:
Overall Officials: Seif E Ahmed, Professor, Study Director — Assiut University
Locations (1):
- Assuit University, Asyut, Egypt

REFERENCES:
- [Background] Maldonado LY, Sergison JE, Gao X, Hubacher D. Menstrual bleeding and spotting with the Levonorgestrel Intrauterine System (52 mg) during the first-year after insertion: a systematic review and meta-analysis. Am J Obstet Gynecol. 2020 May;222(5):451-468.e9. doi: 10.1016/j.ajog.2019.09.044. Epub 2019 Oct 4. PMID 31589865